CLINICAL TRIAL: NCT06042686
Title: Venous Thrombosis Prevention and Sleep Quality: A Comparison of the Kendall and the Recovery Health MAC Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2096
Record Dates: First submitted 2023-08-02; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Deep Venous Thrombosis of Deep Femoral Vein

STUDY DESIGN:
Intervention Model Description: Repeated measures study design where each participant gets both devices on different nights in random order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Repeated measures (Other): Using a 2-day counterbalanced, within-subject repeated-measures design, 16 participants wore two mechanical compression devices, the commonly-used Kendall SCD Express 9525 (SCD) and the novel Recovery Force Movement and Compressions Device (RF-MAC) for 1 night each in their home while sleep was recorded with polysomnography. For each device, participants also completed questionnaires to assess usability, mobility, perceived noise disturbance, and perceived sleep disturbance.
  Interventions: Device: RF Health MAC Device

INTERVENTIONS:
Device: RF Health MAC Device — Using a 2-day counterbalanced, within-subject repeated-measures design, 16 participants wore two mechanical compression devices, the commonly-used Kendall SCD Express 9525 (SCD) and the novel Recovery Force Movement and Compressions Device (RF-MAC) for 1 night each in their home while sleep was recorded with polysomnography. For each device, participants also completed questionnaires to assess usability, mobility, perceived noise disturbance, and perceived sleep disturbance.

SUMMARY:
Venous thromboembolism is prevalent, associated with a high degree of morbidity and mortality, and largely preventable. External mechanical compression is a standard of care for prevention, but compliance with traditional external mechanical compression devices is low due to patient reported issues with comfort, mobility, usability, noise, and sleep disturbances. The purpose of this study was to compare user-rated comfort, mobility, usability, noise, perceived sleep disturbance, and objective sleep disturbance for a novel external lower limb mechanical compression device as compared to a standard sequential compression device.

Using a 2-day counterbalanced, within-subject repeated-measures design, 16 participants wore two mechanical compression devices, the commonly-used Kendall sequential compression device Express 9525 and the novel Recovery Force Movement and Compressions Device for 1 night each in their home while sleep was recorded with polysomnography. For each device, participants also completed questionnaires to assess usability, mobility, perceived noise disturbance, and perceived sleep disturbance.

DETAILED DESCRIPTION:
Recruitment

1. Respondents are solicited via social media/local flyer campaigns (see attached flyers), or word of mouth (see Recruitment via Word of Mouth) to complete a brief, electronic pre-screening survey powered by REDCap software, or to set up a phone call to review study eligibility if preferred.
2. Recruiter responds to eligible or interested Respondents as described in Recruitment Attachments (i.e., Recruitment Email Script).
3. Recruiter coordinates a phone interview with interested and eligible Respondents to confirm eligibility criteria and review the Informed Consent Form with the Respondent in real time over the phone, while the Respondent follows along with a secure REDCap Informed Consent survey to capture an electronic signature.
4. Consenting Participants will submit the Informed Consent form electronically, receive a .pdf copy of their completed (signed) Informed Consent form, and be prompted to complete a subsequent electronic Contact Information Questionnaire, which will only be accessible within the REDCap server by authorized study personnel, e.g. PI and Recruitment Coordinator. A electronic COVID-19 Vaccination Status Confirmation Form will also be completed at this time, including a single upload field for a digital image of the participant's vaccination card. This image will be visually inspected by the Recruiter and immediately deleted from the REDCap server.
5. The Recruiter will manually assign the Participant a coded record ID and follow-up with the Participant via phone or email for tentative scheduling of equipment delivery and data collection through the full protocol. Scheduling will be confirmed with Participants in the week leading up to each transport event.
6. Prior to scheduled data collection, all consenting participants will be screened in their homes for undetected deep vein thrombosis using mobile doppler ultrasound while following all COVID-19 guidelines. Any participant who screens in positive for deep vein thrombosis will be withdrawn from the study.

Study Procedures

1. Once interested respondents have completed all pre-screening, informed consent process will be completed. The voluntary nature of the research will be stressed, participants will have the opportunity to have all of their questions answered, and they will be reminded that they can withdraw their consent at any time.
2. Once consent has been executed and subsequent enrollment forms completed, participants will be scheduled for their deep vein thrombosis screening, their sleep monitoring data collection nights, and their equipment delivery.
3. Participants will then be randomized to receive either the Kendall® or RF Health System on data collection night 1
4. Due to the COVID-19 outbreak, UMass researchers will transport the all study equipment to and from the participants residences using all COVID-19 guidelines and will disinfect all materials at the UMass Sleep Monitoring Laboratory between uses.
5. To ensure high-quality data acquisition, researchers will video conference with participants at prescheduled times, approximately 1-hour prior to participants typical bedtime to provide real-time, remote guidance for proper self-application of the Sleep Profiler headset, Kendall and RF Health System. The first of these sessions will take place shortly after the scheduled deep vein thrombosis screening session. The teleconferencing will take not more of the participant's time than a typical, in-person application.
6. At the conclusion of their first overnight sleep profiler data collection (via Sleep Profiler headset, see attached Technical Manual) while using one of the leg compression devices, participants will be asked to complete their self-report measures in the following order: PROMIS Sleep Disturbance Form 6a, Comfort Rating Scale, Environmental Comfort Scale, System Usability Scale, and Task Load Index.
7. There will be at least one night without any devices between data collection nights 1 & 2.
8. All study procedures will be repeated on data collection overnight 2 using the other external compression device.
9. Once data collection for night 2 has been completed, all participants will be asked if they have any further questions and all questions will be addressed.

ELIGIBILITY:
Inclusion:

* Adult participants age 50-75
* BMI 18-39

Exclusion:

* BMI or age outside of the inclusion criteria limits
* stomach-sleepers
* uncontrolled asthma
* surgery within the past 6 weeks
* history of venous thrombosis within the past 12 months
* abnormalities of the lower extremities, including edema, deformity which does not allow for proper fit of the external mechanical compression devices
* skin breakdown of any kind
* severe peripheral neuropathy
* skin grafting within the last 3 months, cellulitis or dermatitis

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Measure the impact of external mechanical compression on overall sleep. | 4 Months
  Overall sleep will be measured using the Sleep Profiler. The Sleep Profiler is a battery powered portable device that provides a measure of the percentage of overall sleep vs wake in a given period of time.
Compare the comfort associated with mechanical compression between the two devices. | 4 months
  After each night of sleep, participants will provide their self-report on comfort using the Comfort Rating Scale.
Compare the noise associated with mechanical compression between the two devices. | 4 months
  After each night of sleep, participants will provide their self-report on noise using the Environmental Comfort Scale.
Compare the usability associated with mechanical compression between the two devices. | 4 months
  After each night of sleep, participants will provide their self-report on usability using the System Usability Scale.
Compare the perceived sleep disturbance associated with mechanical compression between the two devices. | 4 months
  After each night of sleep, participants will provide their self-report on sleep disturbance using the PROMIS Sleep Disturbance: Short Form 8a.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No